CLINICAL TRIAL: NCT06838832
Title: Novel Allogenic CD19-targeting Chimeric Antigen Receptor γδT Cells Therapy (QH103E) in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Novel Allogenic CD19-targeting CAR-γδT Cell Therapy (QH103E) in r/r NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-091
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: B-cell malignancies; Relapsed or refractory; allogeneic CD19-CAR-γδT; gene editing
MeSH Terms: conditions — Recurrence | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with refractory or relapsed B-cell NHL (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, QH103E product.
  Interventions: Biological: Allogenic CD19-CAR-γδT cell; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Allogenic CD19-CAR-γδT cell — Phase 1 dose escalation (3+3) : dose 1 (1 × 10^6 cells/kg) , dose 2 (3 × 10^6 cells/kg), dose 3 (6× 10^6 cells/kg); Phase 2 : dose of RP2D.
Drug: Fludarabine — Intravenous fludarabine 30~50 mg/m^2/day on days
  -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 500~1000 mg/m^2/ day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
CD19-CAR-γδT cell therapy is a cellular immunotherapy targeting CD19 to perform CAR modification on allogeneic γδT cells. A novel version of the CAR-γδT product by gene editing (QH103E) that has been validated for resistance to alloreactive T cell killing and enhancement of memory efficacy will be used in this study.

This is a single center, prospective, open-label, single-arm, phase 1/2 study. A total of around 30 patients with relapsed or refractory (r/r) B-cell non-Hodgkin's lymphoma (NHL) will be enrolled in the study and receive QH103E product infusion. Phase 1 (n=9 to 12) is dose escalation part, and phase 2 (n=15 to 20) is expansion cohort part. The primary objective of this study was to evaluate the safety and efficacy of QH103E in patients with r/r B-cell NHL.

DETAILED DESCRIPTION:
Phase 1 (dose escalation) In phase 1, 9-12 subjects will be enrolled. Subjects will receive 3 doses of QH103E therapy (1× 10^6 cells/kg; 3× 10^6 cells/kg; 6 × 10^6 cells/kg) increases from low dose to high dose according to the "3 + 3" principle:

1. Three patients were enrolled in the lowest dose group.
2. Subsequent patients were enrolled according to the following rules:

   1. If the incidence of dose limiting toxicity (DLT) was 0/3, 3 patients were enrolled in the next high-dose group.
   2. If the incidence of DLT was 1/3, 3 patients were enrolled at the same dose; If the incidence of DLT was 1/3 + 0/3, 3 patients were enrolled in the next high-dose group. If the incidence of DLT was 1/3 + 1/3, this dose was defined as maximum tolerated dose (MTD); If the incidence of DLT was 1/3 + 2/3 or 1/3 + 3/3, the previous dose was MTD.
   3. If the incidence of DLT was 2/3 or 3/3, the previous dose was MTD. To ensure the safety of the subjects, the first subject in each dose group was observed for at least 28 days after the cell infusion. If no DLT occurred, the remaining two subjects could be enrolled and treated at the same dose level. The safety data of all subjects in each dose group until day 28 should be reviewed and tolerated before proceeding to the next dose group trial. No dose escalation was allowed for the same subject during the trial. If a subject drop out during the observation period due to non-DLT reasons, new subjects should be enrolled to make up for the number of subjects who drop out. Phase 2 (expansion cohort) In phase 2, 15 to 20 subjects will be enrolled and receive QH103E infusion at dose of RP2D, which will be determined based on the MTD, occurrence of DLT, the obtained efficacy results, pharmacokinetics/ pharmacodynamics and other data according to the phase 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. Patients with histologically confirmed CD19-positive B-cell NHL.
3. Relapse after treatment with ≥2 lines systemic therapy for all the B-cell NHL disease types, or refractory disease for aggressive types (DLBCL-NOS, PMBCL, TFL and HGBCL). Relapse disease is defined as disease progression after last regimen. Refractory disease is defined as no CR to first-line therapy:

   * PD as best response to first-line therapy, or
   * SD as best response after at least 4 cycles of first-line therapy (eg,4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy. or refractory post-autologous stem cell transplant (ASCT): i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals); ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.
4. The estimated survival time is over 3 months.
5. The Eastern Cooperative Oncology Group (ECOG) score is 0-2.
6. According to Lugano response criteria 2014, there should be at least one evaluable tumor focus. Evaluable tumor focus was defined as that with the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
7. Subjects must be willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
8. Functions of important organs meet the following requirements:

   Echocardiography showed left ventricular ejection fraction ≥50%. Serum creatinine ≤1.5 × upper limit of normal range (ULN) or endogenous creatinine clearance ≥45mL/min (cockcroft-gault formula); Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤3 times ULN, Total bilirubin ≤1.5× ULN; Pulmonary function: ≤CTCAE grade1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
9. Blood routine (normal values shall not be obtained with growth factors, and hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions below): hemoglobin (Hgb) ≥80g/L, neutrophil count≥1×10^9/L, platelet (PLT) ≥75×10^9/L.
10. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
11. Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
12. No obvious hereditary diseases.
13. Able to understand the requirements and matters of the trial, and willing to participate in clinical research as required.
14. Informed consent must be signed.

Exclusion Criteria:

1. During the screening period, there was central nervous system (CNS) invasion or a history of clinically significant central nervous system diseases, such as epilepsy and cerebrovascular diseases.
2. Women who are pregnant or breastfeeding, or who do not agree to use effective contraception during treatment and during the subsequent 1 year.
3. History of allogeneic hematopoietic stem cell transplantation, or organ transplantation.
4. History of other malignancies that have not been in remission.
5. Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy.
6. Received radiotherapy within 3 months before enrollment.
7. Received immunotherapy drugs within 4 weeks before enrollment, such as anti-programmed death 1 (PD-1) antibody, anti-programmed death ligand 1 (PD-L1) antibody, CD19/CD3-bispecific antibody, and so on.
8. Patients who received any immunocellular therapy within 6 months before enrollment.
9. Confirmed evidence showing positiveness of anti-CD19 scFv reaction in patient serum.
10. Patients who participated in other clinical trials within 4 weeks prior to enrollment.
11. Uncontrolled infectious diseases or other serious illnesses, including but not limited to infections [e.g., human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B (HBV) or C (HCV) infection], congestive heart failure, unstable angina, arrhythmias, or that pose an unpredictable risk in the opinion of the attending physician.
12. The presence of uncontrollable serous membrane fluid, such as massive pleural effusion or ascites.
13. A history of stroke or intracranial hemorrhage within 3 months prior to enrollment.
14. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
15. Received allogeneic cell therapy within 6 weeks prior to enrollment, such as donor lymphocyte infusion.
16. History of allergies to any of the ingredients in cell products.
17. Conditions in which a known mental or physical illness interferes with cooperation with the requirements of the study or disrupts the results or interpretation of the results and, in the opinion of the therapeutic investigator, makes the patient unfit for study participation.
18. There is the situation that the researcher's judgment will interfere with the whole study participation; Situations where there is significant risk to the subject; Or interferes with the interpretation of research data.
19. Inability to understand or unwillingness to sign informed consent.
20. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of lymphodepletion to 12 months after QH103E infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versus-host disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1: Incidence of Dose-Limiting Toxicities (DLTs) | 28 days
  DLT was defined as QH103E-related events with onset within first 28 days following infusion:
  * Grade 3 aGVHD that does not resolve to Grade 1 or 2 within 7 days, with the exception of isolated skin involvement aGVHD;
  * Grade 4 CRS, or grade 3 CRS that does not resolve to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥7 days or Grade 4 ICANS;
  * Any other Grade ≥4 and Grade 3 AE related to the QH103E that lasts for ≥14 days, except hematology toxicity.
Phase 1: Recommended phase 2 dose (RP2D) | 12 months
  The recommended dose for phase 2 was determined through phase 1 study
Phase 2: Best objective Response Rate | 12 months
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as the best response to treatment assessed by investigators and based on the Lugano 2014 assessment criterion.

SECONDARY OUTCOMES:
Phase 2: Overall Survival (OS) | 12 months after the first infusion of QH103E infusion
  OS is defined as the time from QH103E infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 12 months after the first infusion of QH103E infusion
  PFS is defined as the time from the QH103E infusion date to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause. Participants not meeting thecriteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Phase 2: Duration of Response (DOR) | 12 months after the first infusion of QH103E infusion
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B-cell NHL, or death regardless of cause.
Pharmacokinetics: Number and copy number of QH103E (phase 1 and phase 2) | 12 months
  Number and copy number of QH103E were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (QH103E were not detected for two consecutivetimes) to detect the number and copy number of QH103E, and to evaluate the pharmacokinetics of QH103E.
Pharmacodynamics: Peak level of cytokines in serum (phase 1 and phase 2) | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinsese PLA Gereral Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No